CLINICAL TRIAL: NCT05785468
Title: A Retrospective, Observational Study on the Response to Caplacizumab Treatment in aTTP Patients: the Italian Experience (ROSCAPLI)
Acronym: ROSCAPLI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, De Cristofaro Raimondo, Prof. Raimondo De Cristofaro, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4305
Record Dates: First submitted 2023-02-27; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — caplacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Caplacizumab — description and quantification of clinical response in terms of platelet count recovery in patients with aTTP treated t with caplacizumab

SUMMARY:
Thrombotic thrombocytopenic purpura (TTP) is a rare disease with a mortality rate of over 90% if left untreated [1]. TTP is a prototype of the thrombotic microangiopathies (TMAs), and it is characterized by disseminated formation of platelet-rich thrombi in arterioles and capillaries resulting in microangiopathic hemolytic anemia (MAHA), thrombocytopenia, and potential end-organ injury mainly involving the brain, heart, and kidneys leading to significant morbidity/mortality

DETAILED DESCRIPTION:
Thrombotic thrombocytopenic purpura (TTP) is a rare disease with a mortality rate of over 90% if left untreated [1]. TTP is a prototype of the thrombotic microangiopathies (TMAs), and it is characterized by disseminated formation of platelet-rich thrombi in arterioles and capillaries resulting in microangiopathic hemolytic anemia (MAHA), thrombocytopenia, and potential end-organ injury mainly involving the brain, heart, and kidneys leading to significant morbidity/mortality. TTP can either be hereditary or acquired, and the pathogenesis of the latter consists of autoimmune antibodies against the metalloproteinase "a disintegrin and metalloproteinase with a thrombospondin type 1 motif (ADAMTS13)", and ADAMTS13 is responsible for the cleavage of ultra-large multimers of von Willebrand factor (vWF), which induces activation of platelets through glycoprotein Ib-alpha (GPIb-α) receptors and the activated A1 domain of the VWF multimers without a trigger-like endothelial damage or tissue factor. Acquired TTP (aTTP) can be primary (idiopathic) or secondary to some underlying disorders. Therapeutic plasma exchange (PEX) is the mainstay of treatment of aTTP, and with the introduction of PEX, the mortality rate declined dramatically below 20% [1]. The rationale of PEX is the replacement of ADAMTS13, and removal of ultra-large vWF and anti ADAMTS13 antibodies. In newly diagnosed patients with aTTP, PEX and corticosteroids are usually started upfront together [3]. However, a subset of patients may remain refractory to this treatment or have an initial response but relapse after the discontinuation of PEX during the follow-up. There is limited information or consensus available on the management of relapsed/refractory aTTP. While managing PEX refractory patients, PEX may be intensified to 1.5 plasma volume (PV), and even twice daily PEX can be used [4]. In patients remaining refractory to PEX plus corticosteroids, the administration of high-dose methylprednisolone 1 g per day for 3 days can be the choice of treatment [5].Other treatment options in patients with relapsed/refractory TTP may include rituximab, vincristine, cyclophosphamide, cyclosporine A, and splenectomy[6-8]. Caplacizumab is fully reimbursed by the National Health System in Italy since January 2020. While observational data have recently been published in other countries, such as Germany, on the efficacy and safety of caplacizumab [18], cumulative data deriving from the Italian centers that manage the therapy of TTP with caplacizumab have not yet been collected. The aim of this proposal is, therefore,to collect retrospective observationaldata on the response to caplacizumab treatment in patients with aTTP treated with this drug in Italy during the Q4-2019 and Q1-2021.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in this study should have received caplacizumab for treatment in the period between Q4-2019 and the end of February 2021 while the end of follow up observation is scheduled for Q1-2021 (to observe at least one month of post treatment follow up).
* The diagnosis should be based on either clinical/laboratory parameters inclusive of measurement of ADAMTS13 level <10%) or the PLASMIC score (platelets, lysis, active cancer, stem cell or solid organ transplant, MCV, INR, and creatinine) with intermediate and high risk (sore>5) already computed or retrospectively calculated as previously detailed [19] for centers that did not measure the ADAMTS13 level.

Exclusion Criteria:

* Patients treated with uncertain aTTP diagnosis according to the above inclusion criteria - Patients manifesting clinical signs like aTTP but characterized by a different pathogenesis (e.g. cancer, sepsis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a multicenter, retrospective, observational study in patients with aTTP treated with PEX in association with caplacizumab, and immunosuppression between Q4-2019 and 28 February2021.The incidence of aTTP has been estimated at 3-11 cases per million people per year [1-3]. Considering that the adult population of Italy is about 45 million, the number of aTTP cases in Italy is approximately 300 per year. Assuming that 15% of the patients are treated at about 20 sites participating in the study and are eligible to participate, approximately 50 patients can be expected to be included in an 18-month period.The clinical signs will be parametrized by the PLASMIC score and the Glasgow score, where calculated in the various centers. The PLASMIC score and the Glasgow score will be evaluated according to the obtained values (0-4, 5-6, and 7; <13 and 13-15, respectively). All the clinical and laboratory parameters will be taken in each center and reported in the CRF.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
description and quantification of clinical response in terms of platelet count recovery in patients with aTTP treated t with caplacizumab | 18 months
  The primary objective in this study is the description of clinical response in terms of platelet count recovery in patients with aTTP treated with caplacizumab , in addition to PEX and immunosuppression in the real-world setting.
The primary objective in this study is the quantification of clinical response in terms of platelet count recovery in patients with aTTP treated t with caplacizumab | 18 months
  The primary objective in this study is the quantification of clinical response in terms of platelet count recovery in patients with aTTP treated with caplacizumab , in addition to PEX and immunosuppression in the real-world setting.

SECONDARY OUTCOMES:
evaluation of number of exacerbations,rate of relapse and TTP-related mortality | 18 months
  Secondary objectives include:
  a) Number of exacerbations, defined as recurrent thrombocytopenia within 30 days after the end of therapy;
evaluation of number of exacerbations,rate of relapse and TTP-related mortality | 18 months
  Secondary objectives include:
  b) Rate of relapse, defined as a TTP event occurring more than 30 days after the end of daily plasma exchange;
evaluation of number of exacerbations,rate of relapse and TTP-related mortality | 18 months
  Secondary objectives include:
  c) Refractoriness; defined by the lack of a doubling of platelet count after 4 days of treatment and a lactate dehydrogenase level that remained above the upper limit of the normal range
evaluation of number of exacerbations,rate of relapse and TTP-related mortality | 18 months
  Secondary objectives include:
  d) TTP-related mortality
evaluation of number of exacerbations,rate of relapse and TTP-related mortality | 18 months
  Secondary objectives include:
  e) Evaluation of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- FPG, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided